CLINICAL TRIAL: NCT00896571
Title: Single-center,Open-label, Uncontrolled Study to Investigate the Effects of the Transdermal Contraceptive Patch Containing 0.55 mg Ethinylestradiol and 2.1 mg Gestodene on the Endometrium in a 21-day Regimen for 13 Cycles in 80 Healthy Women
Brief Title: Transdermal Contraceptive Patch - Endometrial Effects Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14287; 2009-010599-45 (EudraCT Number)
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Contraception
Keywords: Fertility control; Contraception
MeSH Terms: interventions — Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestogene (BAY86-5016)

INTERVENTIONS:
Drug: Ethinylestradiol/Gestogene (BAY86-5016) — 7-day patch containing 0.55 mg ethinylestradiol (EE) and 2.1 mg gestodene (GSD) in a 21-day regimen

SUMMARY:
The aim of the present study is to investigate the effects of the transdermal patch on the endometrium in healthy women who require contraception.

ELIGIBILITY:
Inclusion Criteria:

* Requiring contraception
* Normal cervical smear
* Smokers not older than 30 years
* History of regular cyclic menstrual periods

Exclusion Criteria:

* Pregnancy or lactation
* Obesity (BMI> 30 kg/m2)
* Significant skin reaction to transdermal preparations or sensitivity to surgical / medical tape
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Use of other contraceptive methods than study medication

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Effect on the endometrium at cycle 13 | 13 treatment cycles (each consisting of 28 days)

SECONDARY OUTCOMES:
Cervical smear | 13 treatment cycles (each consisting of 28 days)
Adverse events | 13 treatment cycles (each consisting of 28 days)
Cycle control | 13 treatment cycles (each consisting of 28 days)
Safety laboratory | 13 treatment cycles (each consisting of 28 days)
Occurence of pregnancy | 13 treatment cycles (each consisting of 28 days)

OTHER OUTCOMES:
Treatment compliance | 13 treatment cycles (each consisting of 28 days)
Subjective assessment of satisfaction with the treatment | 13 treatment cycles (each consisting of 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- See also: Click here and search for EMA websynopsis result — http://www.clinicaltrialsregister.eu